CLINICAL TRIAL: NCT04853862
Title: Quality of Life Assessment Study in Patients With Metastatic Head and Neck Neoplasia Submitted to Immunotherapy in Brazil
Brief Title: Quality of Life in Head and Neck Patients
Acronym: QLiHN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcos Santos, MD PhD, University of Brasilia
Other Study IDs: CONFIAR
Record Dates: First submitted 2021-04-17; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Cancer
Keywords: head and neck; immunotherapy; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Questionnaire for health-related quality of life evaluation
  Other Names: EORTC H&N-43

SUMMARY:
Evaluation of health-related quality of life of head and neck cancer patients undergoing immunotherapy

DETAILED DESCRIPTION:
Introduction: The treatment of head and neck neoplasms, as well as the evolution of the disease, can affect a variety of body functions, including breathing, swallowing and speech, with great potential to cause various physical, emotional, and social problems to the patient, leading to considerable impairment of their quality of life. Several instruments were developed to measure this variable. Such evaluation is currently considered fundamental to report therapeutic results, but there is no consensus regarding the instrument to be employed. The University of Washington questionnaire has been the most widely used so far. EORTC (European Organization for Cancer Research and Treatment) recently published a new questionnaire specifically for patients treated for head and neck cancer (EORTC QLQ-H & N43), already validated in Portuguese for Brazil.

Objectives: The aim of this prospective and multi-institutional study is to evaluate the quality of life of patients with metastatic head and neck cancer undergoing immunotherapy in different regions of Brazil. Other endpoints will also be evaluated such as disease-free survival and overall survival.

Procedures: EORTC QLQ-30 and EORTC QLQ-H & N43 questionnaires, validated in Portuguese for Brazil, will be applied to all patients with metastatic head and neck neoplasms undergoing immunotherapy at participating institutions. These will be evaluated before the beginning of the treatment and then every 2 months, for an estimated period of 2 years or until death or on demand, in case of symptomatology that justifies it.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of recurrent or metastatic squamous cell carcinoma of the head and neck region, whose planned treatment is immunotherapy, will be included. We will consider, separately, patients that had been treated with platinum before (platinum-refractory) and patients that were not submitted to this treatment (platinum naïve).

Primary site: patients with primary pharyngeal tumors (oro or hypopharynx), oral cavity and larynx will be included.

Exclusion Criteria:

* Patients with cognitive impairment that prevents the proper application of questionnaires
* Brain metastasis
* Autoimmune disease
* Systemic immunosuppressive treatment
* Hepatitis B, C or HIV infection
* Prior immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients undergoing systemic treatment with immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 2 years
  Evaluation of quality of life based on validated questionnaire
Overall survival | 2 years
  Overall survival

IPD SHARING:
Plan to Share IPD: Yes
Data base will be shared, if requested
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available from December 2023 to December 2028
Access Criteria: Request by email